CLINICAL TRIAL: NCT05091918
Title: FS5 Limited Market Release - MotionSense Clinical Use Evaluation
Brief Title: Limited Market Release - MotionSense Clinical Use Evaluation
Acronym: FS5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orthosensor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Orthosensor
Record Dates: First submitted 2021-10-13; First posted 2021-10-25 (Actual); Results first posted 2023-09-07 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-06

CONDITIONS: Knee Arthroplasty; Patient Engagement; Patient-Reported Outcome Measures (PROMs)
Keywords: MotionSense
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- MotionSense Wearable (Other): Using MotionSense from pre-op to 90 days post-op during the recovery after primary TKA
  Interventions: Device: MotionSense

INTERVENTIONS:
Device: MotionSense — MotionSense Wearable: Remote patient monitoring

SUMMARY:
Prospective evaluation of patient compliance and prescribed home exercise program using MotionSense wearable system during recovery from primary total knee arthroplasty.

DETAILED DESCRIPTION:
During the proposed study, the MotionSense wearable system will be used by patients undergoing total knee arthroplasty (TKA) surgery leading up to and after their surgery. The patients will be using the system to monitor their recovery during daily activities, log daily pain scores and patient reported outcomes while also supporting their prescribed home exercise program. Each patient will thereby participate in outpatient physiotherapy in line with their current standard of care, while the physiotherapist will leverage the opportunities of the presented platform to give the patient personalized reminders for their patient-specific home exercise program. The surgeon / research nurse will additionally be able to monitor the patients recovery remotely as the sensor / app data is shared to the OrthoLogIQ platform.

ELIGIBILITY:
Inclusion Criteria:

* Planned for unilateral total knee surgery in the coming 4 weeks
* Age 50 to 80
* Owns a smart phone

Exclusion Criteria:

* BMI exceeding 35
* Severe skin conditions

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Oklahoma Joint Reconstruction Institute, Oklahoma City, Oklahoma
  - Robotic Joint Replacement Institute LLC, Wakefield, Rhode Island

RESULTS

PARTICIPANT FLOW:
Groups:
- Motionsense Wearable Group: Using Motionsense from pre-op to 90 days post-op during the recovery after primary TKA
  Motionsense Wearable: Remote patient monitoring
Period: Overall Study
Arm/Group | Motionsense Wearable Group
Started | 101
Completed | 19
Not Completed | 82
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 81

BASELINE CHARACTERISTICS:
Groups:
- Motionsense Wearable Group: Using Motionsense from up to 30 days pre-op and 90 days post-op during the recovery after primary TKA
  Motionsense Wearable: Remote patient monitoring
Arm/Group | Motionsense Wearable Group
Number analyzed (Participants) | 101
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [60 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic | 3
  Ethnicity: Native | 1
  Ethnicity: White | 80
  Ethnicity: Other/Multiple | 3
  Ethnicity: Declined to respond | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 101

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Patient and Practice Compliance With the MotionSense Wearable System: Hours of MotionSense Use Per Day in Office
Description: Hours spent per day in office by practice using MotionSense wearable system, from 30 days preoperative to 90 days postoperative.
Time Frame: 30 days preoperative to 90 days postoperative
Population: The office staff did not collect data on the hours spent per day in office, except for onboarding time, which is Outcome Measure 5.
Groups:
- MotionSense Wearable Group: Using MotionSense from pre-op to 90 days post-op during the recovery after primary TKA
Arm/Group | MotionSense Wearable Group
Number analyzed (Participants) | 0

2. Primary Outcome: Evaluate Patient and Practice Compliance With the MotionSense Wearable System: Number of Days Use After / Prior to Surgery
Description: Initial and last day worn while wearing MotionSense from 30 days preoperative to 90 days postoperative
Time Frame: 30 days preoperative to 90 days postoperative
Population: Preoperative participants: 2 Patients did not wear device preoperatively. Postoperative participants: 23 Patients did not wear device postoperatively.
Measure: Median (Inter-Quartile Range); unit: Days relative to surgery
Arm/Group | MotionSense Wearable Group
Number analyzed (Participants) | 101
Days relative to surgery
  Preoperative day of initial use: number analyzed (Participants) | 99
  Preoperative day of initial use | -12 [-14 to -7]
  Preoperative day of last use: number analyzed (Participants) | 99
  Preoperative day of last use | -1 [-4 to -1]
  Postoperative day of initial use: number analyzed (Participants) | 78
  Postoperative day of initial use | 2 [1 to 5]
  Postoperative day of last use: number analyzed (Participants) | 78
  Postoperative day of last use | 68 [36 to 89]

3. Primary Outcome: Evaluate Patient and Practice Compliance With the MotionSense Wearable System: Filled Out Questionnaires
Description: Count of participants who have completed the aggregate questionnaires in the MotionSense App downloaded to their mobile devices at each timepoint for evaluation of compliance with the MotionSense Wearable System.
Time Frame: Preoperative, 2 weeks postoperative, 6 weeks postoperative, 90 days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | MotionSense Wearable Group
Number analyzed (Participants) | 101
Participants
  Preoperative questionnaire | 87
  Postoperative 2 week questionnaire | 58
  Postoperative 6 week questionnaire | 50
  Postoperative 90 day questionnaire | 15

4. Primary Outcome: Evaluate Patient and Practice Compliance With the MotionSense Wearable System: Home Exercise Program
Description: Percent of exercise sessions completed while wearing MotionSense from 30 days preoperative to 90 days postoperative.
  An exercise session is a collection of exercises that can be customized and assigned to a patient to be performed either once or twice a day.
Time Frame: 30 days preoperative to 90 days postoperative
Population: There were 10 patients who did not have any exercise data that was completed.
Measure: Median (Inter-Quartile Range); unit: Percent of completed exercise sessions
Arm/Group | MotionSense Wearable Group
Number analyzed (Participants) | 91
Percent of completed exercise sessions | 19 [6 to 40]

5. Primary Outcome: Evaluate Patient and Practice Compliance With the MotionSense Wearable System: Patient Onboarding Time in Surgeon Clinic
Description: Minutes spent per patient at preoperative onboarding visit. Onboarding visit provided patients with instructions on system use and initial wearable installation.
Time Frame: Preoperative onboarding visit
Population: There were 7 patients who did not have onboarding time data collected.
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | MotionSense Wearable Group
Number analyzed (Participants) | 94
Minutes | 32 [25 to 42]

6. Primary Outcome: Document Home Exercise Program Prescribed to Patients Throughout Their Individualized Recovery Progress by Surgeons and Physiotherapists
Description: Daily percentage of patients prescribed each home exercise during preoperative, 1-30 days postoperative, 31-60 days postoperative, 61-90 days postoperative time periods.
  Isometric quads: Lie back to floor, tense quadriceps, hold, repeat. Sit-to-stands: Sit, stand, strengthen, repeat. Short-arc quadriceps: Lie back to floor with leg bent, extend leg, hold, repeat.
  Heel slides: Lie back to floor, slide and bend leg, hold, repeat. Hamstring curls: Lie stomach to floor, bend leg, hold, repeat. Long-arc quadriceps: Sit, lift, hold, count, repeat, strengthen. Straight leg raises: Lie back to floor, lift leg, hold, lower, repeat. Standing knee bends: Stand, squat, knees, lower, maintain form, repeat. Knee straightening stretches: Lie back to floor, extend leg, tense, relax. Sitting knee bends: Sit, hold, stretch, hold, slide, repeat. Assisted knee stretches: Sit, bend, hold, release, repeat. Warmup: 5 minutes
Time Frame: Preoperative, 1-30 days postoperative, 31-60 days postoperative, 61-90 days postoperative
Measure: Median (Inter-Quartile Range); unit: Percent of participants assigned
Arm/Group | MotionSense Wearable Group
Number analyzed (Participants) | 101
Percent of participants assigned
  Pre-op: Isometric quads | 22 [5 to 68]
  Pre-op: Sit-to-stands | 0 [0 to 0]
  Pre-op: Short-arc quads | 22 [5 to 68]
  Pre-op: Heel slides | 21 [4 to 67]
  Pre-op: Hamstring curls | 0 [0 to 0]
  Pre-op: Long-arc quads | 0 [0 to 0]
  Pre-op: Straight-leg raises | 1 [1 to 2]
  Pre-op: Standing knee bends | 0 [0 to 0]
  Pre-op: Knee straightening stretches | 22 [5 to 68]
  Pre-op: Sitting knee bends | 0 [0 to 0]
  Pre-op: Assisted knee stretches | 1 [1 to 1]
  Pre-op: Warmup | 22 [5 to 68]
  0-30 days post-op: Isometric quads | 87 [85 to 91]
  0-30 days post-op: Sit-to-stands | 2 [0 to 9]
  0-30 days post-op: Short-arc quads | 85 [82 to 91]
  0-30 days post-op: Heel slides | 87 [85 to 90]
  0-30 days post-op: Hamstring curls | 0 [0 to 0]
  0-30 days post-op: Long-arc quads | 11 [5 to 20]
  0-30 days post-op: Straight-leg raises | 10 [6 to 20]
  0-30 days post-op: Standing knee bends | 8 [3 to 18]
  0-30 days post-op: Knee straightening | 87 [82 to 91]
  0-30 days post-op: Sitting knee bends | 7 [4 to 13]
  0-30 days post-op: Assisted knee stretches | 4 [3 to 7]
  0-30 days post-op: Warm | 87 [83 to 91]
  31-60 days post-op: Isometric quads | 65 [61 to 70]
  31-60 days post-op: Sit-to-stands | 24 [20 to 26]
  31-60 days post-op: Short-arc quads | 66 [62 to 70]
  31-60 days post-op: Heel slides | 72 [69 to 74]
  31-60 days post-op: Hamstring curls | 11 [7 to 14]
  31-60 days post-op: Long-arc quads | 28 [26 to 28]
  31-60 days post-op: Straight-leg raises | 31 [29 to 31]
  31-60 days post-op: Standing knee bends | 28 [26 to 28]
  31-60 days post-op: Knee straightening | 65 [63 to 70]
  31-60 days post-op: Sitting knee bends | 22 [19 to 22]
  31-60 days post-op: Assisted knee stretches | 16 [14 to 16]
  31-60 days post-op: Warmup | 73 [72 to 75]
  61-90 days post-op: Isometric quads | 55 [53 to 57]
  61-90 days post-op: Sit-to-stands | 29 [29 to 30]
  61-90 days post-op: Short-arc quads | 56 [54 to 58]
  61-90 days post-op: Heel slides | 64 [62 to 65]
  61-90 days post-op: Hamstring curls | 17 [16 to 17]
  61-90 days post-op: Long-arc quads | 28 [28 to 30]
  61-90 days post-op: Straight-leg raises | 29 [28 to 30]
  61-90 days post-op: Standing knee bends | 27 [26 to 27]
  61-90 days post-op: Knee straightening | 57 [55 to 58]
  61-90 days post-op: Sitting knee bends | 21 [21 to 21]
  Assisted knee stretches | 16 [16 to 16]
  61-90 days post-op: Warmup | 67 [65 to 67]

7. Secondary Outcome: Correlate Functional and Patient Reported Outcome Metrics
Description: Spearman correlation of mean step count to Knee Injury and Osteoarthritis Outcome Score (KOOS) patient questionnaire.
  The Statistical Spearman correlation coefficient evaluates relationships between variables. The Spearman correlation coefficient is used to evaluate the relationship of the mean step count to the Knee Injury and Osteoarthritis Outcome Score (KOOS) patient questionnaire. The KOOS consists of 5 subscales: Pain, other symptoms, function in daily living (ADL), function in sport and recreation and knee related quality of life (QOL).
  The Spearman Correlation coefficients range from -1to 1. If r = 0, there is no linear relationship between the variables. If r=+1, there is a strong direct relationship. If r = -1, there is a strong inverse relationship.
Time Frame: 2 weeks, 6 weeks, 90 days postoperative
Population: At 2 weeks (-5 days), 60 patients did not have completed data for KOOS or step count.
  At 6 weeks (-5 days), 61 patients did not have completed data for KOOS or step count.
  At 90 days (-5 days), 90 patients did not have completed data for KOOS or step count.
Measure: Number; unit: Spearman Correlation Coefficient
Arm/Group | MotionSense Wearable Group
Number analyzed (Participants) | 101
Spearman Correlation Coefficient
  KOOS: ADL, 2 weeks: number analyzed (Participants) | 41
  KOOS: ADL, 2 weeks | 0.24
  KOOS: ADL, 6 weeks: number analyzed (Participants) | 40
  KOOS: ADL, 6 weeks | 0.21
  KOOS: ADL, 90 days: number analyzed (Participants) | 11
  KOOS: ADL, 90 days | -0.01
  KOOS: Pain, 2 weeks: number analyzed (Participants) | 41
  KOOS: Pain, 2 weeks | 0.07
  KOOS: Pain, 6 weeks: number analyzed (Participants) | 40
  KOOS: Pain, 6 weeks | 0.21
  KOOS: Pain, 90 days: number analyzed (Participants) | 11
  KOOS: Pain, 90 days | 0.17
  KOOS: QoL, 2 weeks: number analyzed (Participants) | 41
  KOOS: QoL, 2 weeks | 0.16
  KOOS: QoL, 6 weeks: number analyzed (Participants) | 40
  KOOS: QoL, 6 weeks | 0.11
  KOOS: QoL, 90 days: number analyzed (Participants) | 11
  KOOS: QoL, 90 days | 0.09
  KOOS: Sport/Recreation, 2 weeks: number analyzed (Participants) | 41
  KOOS: Sport/Recreation, 2 weeks | 0.08
  KOOS: Sport/Recreation, 6 weeks: number analyzed (Participants) | 40
  KOOS: Sport/Recreation, 6 weeks | 0.01
  KOOS: Sport/Recreation, 90 days: number analyzed (Participants) | 11
  KOOS: Sport/Recreation, 90 days | 0.16
  KOOS: Symptoms, 2 weeks: number analyzed (Participants) | 41
  KOOS: Symptoms, 2 weeks | 0.12
  KOOS: Symptoms, 6 weeks: number analyzed (Participants) | 40
  KOOS: Symptoms, 6 weeks | -0.02
  KOOS: Symptoms, 90 days: number analyzed (Participants) | 11
  KOOS: Symptoms, 90 days | -0.23

8. Secondary Outcome: Evaluate Convenience of Using the MotionSense System: Number of Leg Registrations Performed (Per Day)
Description: Number of leg registrations performed (per day) per patient, while wearing MotionSense from 30 days preoperative to 90 days postoperative.
Time Frame: 30 days preoperative to 90 days postoperative
Population: The number of leg registrations performed per day per patient was not collected. These data collections were not technically feasible.
Arm/Group | Motionsense Wearable Group
Number analyzed (Participants) | 0

9. Secondary Outcome: Evaluate Convenience of Using the MotionSense System: Number of (Weekly / Daily) Patches Used
Description: Number of weekly and daily patches used per patient, while wearing MotionSense from 30 days preoperative to 90 days postoperative.
Time Frame: 30 days preoperative to 90 days postoperative
Population: The number of weekly and daily patches used per patient was not collected. Accurate data collection was unattainable by office staff.
Arm/Group | Motionsense Wearable Group
Number analyzed (Participants) | 0

10. Secondary Outcome: Evaluate Convenience of Using the MotionSense System: Number of Wound Pictures Shared With Surgeon Office
Description: Total number of wound pictures shared with surgeon office per patient while wearing MotionSense from 30 days preoperative to 90 days postoperative
Time Frame: 30 days preoperative to 90 days postoperative
Measure: Mean (Inter-Quartile Range); unit: Shared pictures
Arm/Group | MotionSense Wearable Group
Number analyzed (Participants) | 101
Shared pictures | 7 [0 to 17]

11. Secondary Outcome: Establish Normative Recovery Data for the Primary Outcome Metrics Captured by the MotionSense System: Daily VAS Pain Scores
Description: Visual Analog Scale (VAS) pain scores while wearing MotionSense from 30 days preoperative to 90 days postoperative
  The VAS pain score is a patient questionnaire to assess the subjective pain intensity. The VAS is a horizontal line ranging from 0 to 10, where 0 represents no pain and 10 represents the worst possible pain.
Time Frame: 30 days preoperative to 90 days postoperative
Population: 4 patients were not included in the analysis because they did not produce pain scores.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | MotionSense Wearable Group
Number analyzed (Participants) | 97
units on a scale | 3 [2 to 4]

12. Secondary Outcome: Establish Normative Recovery Data for the Primary Outcome Metrics Captured by the MotionSense System: Daily Steps
Description: Daily steps while wearing MotionSense from 30 days preoperative to 90 days postoperative
Time Frame: 30 days preoperative to 90 days postoperative
Population: There were 4 patients who did not produce daily steps or wear device for longer than 10 minutes per day.
Measure: Median (Inter-Quartile Range); unit: Daily steps
Arm/Group | MotionSense Wearable Group
Number analyzed (Participants) | 97
Daily steps | 2519 [886 to 4771]

13. Secondary Outcome: Establish Normative Recovery Data for the Primary Outcome Metrics Captured by the MotionSense System: Knee Active and Weight Bearing Time
Description: Scores while wearing MotionSense from 30 days preoperative to 90 days postoperative
  Knee active time is the time the patient spends moving the knee per day. Weight bearing time is the time the patient spends with the leg in an upright position per day.
Time Frame: 30 days preoperative to 90 days postoperative
Population: There were 4 patients who did not produce knee active or weight bearing time, or wear the device for greater than 10 minutes per day.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | MotionSense Wearable Group
Number analyzed (Participants) | 101
minutes
  Weight bearing time | 142 [82 to 214]
  Knee active time | 60 [32 to 94]

14. Secondary Outcome: Establish Normative Recovery Data for the Primary Outcome Metrics Captured by the MotionSense System: Range of Motion
Description: Scores while wearing MotionSense from 30 days preoperative to 90 days postoperative
  Range of Motion (ROM) for the knee refers to the degree of movement that can be achieved at the knee joint. It describes the arc or extent of motion from full extension (straightening) to full flexion (bending) in degrees.
Time Frame: 30 days preoperative to 90 days postoperative
Population: There were 12 patients who did not produce ROM data, wear the device for long enough (>10 mins/day), or were excluded due to data quality concerns.
Measure: Median (Inter-Quartile Range); unit: Degrees
Arm/Group | MotionSense Wearable Group
Number analyzed (Participants) | 89
Degrees | 110 [100 to 120]

15. Secondary Outcome: Establish Normative Recovery Data for the Primary Outcome Metrics Captured by the MotionSense System: Gait Quality (Steps Per Minute)
Description: Steps per minute while wearing MotionSense from 30 days preoperative to 90 days postoperative
Time Frame: 30 days preoperative to 90 days postoperative
Population: Gait analysis was incomplete for 16 patients.
Measure: Median (Inter-Quartile Range); unit: Steps per minute
Arm/Group | MotionSense Wearable Group
Number analyzed (Participants) | 85
Steps per minute | 47 [42 to 52]

ADVERSE EVENTS:
Time Frame: 30 days pre-op until 90 days post-op
Arm/Group | Motionsense Wearable Group
All-Cause Mortality (participants affected / at risk) | 0/101
Serious Adverse Events (participants affected / at risk) | 2/101
Other Adverse Events (participants affected / at risk) | 10/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Motionsense Wearable Group (N=101)
Deep joint infection (Infections and infestations) | 1 — Bacterial infection was the result of a plastic surgery. Source was plastic surgery, not the total knee SURGERY.
Knee stiffness Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 1 — Pain and stiffness requiring manipulation under anesthesia
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Motionsense Wearable Group (N=101)
Skin reaction (Skin and subcutaneous tissue disorders) | 10

LIMITATIONS AND CAVEATS:
Comment for Document Section: Initially the Ethical Review Committee did not request a detailed Statistical Analysis Plan. The Statistical Analysis Plan was uploaded to describe the standard analysis for descriptive statics. The study concluded on August 1, 2022. Therefore, belated IRB approval of the standard statistical analysis plan was not requested.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/18/NCT05091918/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-18): https://cdn.clinicaltrials.gov/large-docs/18/NCT05091918/SAP_001.pdf